CLINICAL TRIAL: NCT06897683
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSES OF CARBAMAZEPINE ON THE PHARMACOKINETICS OF SINGLE DOSE PF-07220060 ADMINISTERED UNDER THE FED CONDITION TO HEALTHY PARTICIPANTS
Brief Title: A Study to Learn if the Study Medicine Called Carbamazepine Changes How the Body Processes PF-07220060
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4391012
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adults
Keywords: PF-07220060; Carbamazepine; Drug-drug interaction

STUDY DESIGN:
Intervention Model Description: This is an open-label, fixed sequence, two-period, crossover study in healthy participants.
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): Single dose PF-07220060 alone
  Interventions: Drug: PF-07220060
- Period 2 (Experimental): Single dose PF-07220060 given after multiple doses of carbamazepine
  Interventions: Drug: PF-07220060; Drug: Carbamazepine ER Tablet

INTERVENTIONS:
Drug: PF-07220060 — Single dose PF-07220060 tablet administered with a moderate-fat standard calorie meal
Drug: Carbamazepine ER Tablet — Carbamazepine dosing titration regimen in Period 2 from Day 1 to 18
  Arms: Period 2

SUMMARY:
The purpose of this study is to learn how carbamazepine changes how the body processes PF-07220060 in the body of healthy adults.

This study will happen in 2 periods. The purpose of Period 1 of the study is to understand how the medicine is changed and eliminated from the body after it is taken) and safety of a single dose of PF-07220060.

The purpose of Period 2 of the study is to understand how the medicine is changed and eliminated from the body after it is taken and safety of a single dose of PF-07220060 following multiple days dosing carbamazepine twice a day.

Multiple blood samples will be collected in each period up to 120 hours after the PF-07220060 dose in order to measure the amount of PF-07220060 in the blood. On Day 1 in Period 1, a single oral dose of PF-07220060 will be administered with food. Period 2 will begin following the last blood sample collection in Period 1. Carbamazepine will be dosed in Period 2 at 100 mg twice a day on Days 1, 2, and 3, and then, will increase to 200 mg twice a day on Days 4, 5, 6, and 7, and will eventually increase to and be maintained at 300 mg twice a day for the rest of Period 2 from Day 8 to Day 18. On Day 14 in Period 2, a single oral dose of PF-07220060 will be administered.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants aged 18 to 65 years at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Body mass index (BMI) of 17.5-30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Evidence of a personally signed and dated ICD indicating that the participant has been informed of all pertinent aspects of the study.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

Key Exclusion Criteria:

* Participants shown to carry or be positive for human leukocyte antigen (HLA)-B*1502 and HLA-A*3101 (genotyping alleles/markers related with carbamazepine-associated SJS or TEN).
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Concomitant use of any medications or substances that are strong inducers or inhibitors of CYP3A4 or UGT2B7 are prohibited within 5 half-lives plus 14 days (up to 56 days) prior to first dose of PF 07220060.
* Previous administration with a study intervention (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* History of sensitivity to carbamazepine, tricyclic compounds, or any of the formulation components of carbamazepine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-05-11 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Plasma PF-07220060 Maximum Observed Plasma Concentration (Cmax) | Pre-dose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose.
Plasma PF-07220060 Area under the plasma concentration versus time curve (AUC) | Pre-dose, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose.

SECONDARY OUTCOMES:
Number of Participants With Laboratory Abnormalities | From baseline up to 28 to 35 days after last dose of investigational drug
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings | From baseline up to 28 to 35 days after last dose of investigational drug
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | From baseline up to 28 to 35 days after last dose of investigational drug
Number of Participants With Treatment-Emergent Adverse Events (AEs) | From baseline up to 28 to 35 days after last dose of investigational drug

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391012